CLINICAL TRIAL: NCT03070782
Title: A Randomized, Double-blind, Placebo-Controlled, Dose-Ranging Phase 2 Study of ISIS 681257 (AKCEA-APO(a)-LRx) Administered Subcutaneously to Patients With Hyperlipoproteinemia(a) and Established Cardiovascular Disease (CVD)
Brief Title: Phase 2 Study of ISIS 681257 (AKCEA-APO(a)-LRx) in Participants With Hyperlipoproteinemia(a) and Cardiovascular Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akcea Therapeutics (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISIS 681257-CS6; 2016-003373-18 (EudraCT Number)
Record Dates: First submitted 2017-01-31; First posted 2017-03-06 (Actual); Results first posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Elevated Lipoprotein(a); Cardiovascular Disease
Keywords: IONIS-APO(a)-LRx; AKCEA-APO(a)-LRx; Dyslipidemia; Dyslipoproteinemia; Hyperlipidemia; Hyperlipoproteinemia; Hyperlipoproteinemia(a); Hyperlipoproteinemia a; Lipoprotein; Lipoprotein(a); Lipoprotein a; Lp(a); Lp a
MeSH Terms: conditions — Cardiovascular Diseases; Dyslipidemias; Hyperlipidemias; Hyperlipoproteinemias | interventions — AKCEA-APO(a)-LRx; pelacarsen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort A: ISIS 681257: 20 mg Q4W (Experimental): Cohort A participants received 20 milligrams (mg) ISIS 681257, subcutaneous (SC) injection, once every 4 weeks (Q4W), for up to 49 weeks and a maximum of 13 doses.
  Interventions: Drug: ISIS 681257
- Cohort B: ISIS 681257: 40 mg Q4W (Experimental): Cohort B participants received 40 mg of ISIS 681257, SC injection, once Q4W, for up to 49 weeks and a maximum of 13 doses.
  Interventions: Drug: ISIS 681257
- Cohort C: ISIS 681257: 60 mg Q4W (Experimental): Cohort C participants received 60 mg of ISIS 681257, SC injection, once Q4W, for up to 49 weeks and a maximum of 13 doses.
  Interventions: Drug: ISIS 681257
- Cohort D: ISIS 681257: 20 mg Q2W (Experimental): Cohort D participants received 20 mg of ISIS 681257, SC injection, once every 2 weeks (Q2W), for up to 51 weeks and a maximum of 26 doses.
  Interventions: Drug: ISIS 681257
- Cohort E: ISIS 681257: 20 mg QW (Experimental): Cohort E participants received 20 mg of ISIS 681257, SC injection, once weekly (QW), for up to 52 weeks and a maximum of 52 doses.
  Interventions: Drug: ISIS 681257
- Placebo (Placebo Comparator): Participants in each cohort were randomized to receive placebo at a dose-matched volume of study drug (ISIS 681257).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ISIS 681257 — ISIS 681257 solution for SC injection.
  Other Names: AKCEA-APO(a)-LRx, IONIS-APO(a)-LRx, TQJ230 and Pelacarsen
  Arms: Cohort A: ISIS 681257: 20 mg Q4W; Cohort B: ISIS 681257: 40 mg Q4W; Cohort C: ISIS 681257: 60 mg Q4W; Cohort D: ISIS 681257: 20 mg Q2W; Cohort E: ISIS 681257: 20 mg QW
Drug: Placebo — Sterile normal saline (0.9% NaCl)
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, dose-ranging study to evaluate the safety, including tolerability, of ISIS 681257 and to assess the efficacy of different doses and dosing regimens of ISIS 681257 for reduction of plasma Lipoprotein(a) [Lp(a)] levels in participants with hyperlipoproteinemia(a) and established cardiovascular disease (CVD).

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of CVD defined as documented coronary artery disease, stroke, or peripheral artery disease
* Lp(a) plasma level ≥ 60 mg/dL
* Must be on standard-of-care preventative therapy for other than elevated Lp(a) CVD risk factors

Key Exclusion Criteria:

* Within 6 months of Screening: acute coronary syndrome, major cardiac surgery, or stroke/TIA
* Within 3 months of Screening: coronary, carotid, or peripheral arterial revascularization, major non-cardiac surgery, or lipoprotein apheresis
* Heart failure New York Heart Association (NYHA) class IV

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-11-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (21):
  - Clinical Site, Cottonwood, Arizona
  - Clinical Site, Huntington Beach, California
  - Clinical Site, La Jolla, California
  - Clinical Site, Los Angeles, California
  - Clinical Site, Stanford, California
  - Clinical Site, Colorado Springs, Colorado
  - Clinical Site, Boca Raton, Florida
  - Clinical Site, Jacksonville, Florida
  - Clinical Site, Kansas City, Kansas
  - Clinical Site, Baltimore, Maryland
  - Clinical Site, Boston, Massachusetts
  - Clinical Site, Cooperstown, New York
  - Clinical Site, New York, New York
  - Clinical Site, Cleveland, Ohio
  - Clinical Site, Portland, Oregon
  - Clinical Site, Lancaster, Pennsylvania
  - Clinical Site, Philadelphia, Pennsylvania
  - Clinical Site, Providence, Rhode Island
  - Clinical Site, Houston, Texas
  - Clinical Site, Falls Church, Virginia
  - Clinical Site, Milwaukee, Wisconsin
- Canada (4):
  - Clinical Site, Chicoutimi, Quebec
  - Clinical Site, Montreal, Quebec
  - Clinical Site, Québec, Quebec
  - Clinical Site, Ottawa
- Denmark (2):
  - Clinical Site, Herlev
  - Clinical Site, Viborg
- Germany (2):
  - Clinical Site, Berlin
  - Clinical Site, Cologne
- Clinical Site, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tekendo-Ngongang C, Gleeson JG, Mignon L. Treating the Untreatable: Antisense Oligonucleotides as an Individualized Therapy for Rare Genetic Kidney Diseases. J Am Soc Nephrol. 2024 Dec 1;35(12):1774-1777. doi: 10.1681/ASN.0000000532. Epub 2024 Sep 27. No abstract available. PMID 39331470
- [Derived] Stiekema LCA, Prange KHM, Hoogeveen RM, Verweij SL, Kroon J, Schnitzler JG, Dzobo KE, Cupido AJ, Tsimikas S, Stroes ESG, de Winther MPJ, Bahjat M. Potent lipoprotein(a) lowering following apolipoprotein(a) antisense treatment reduces the pro-inflammatory activation of circulating monocytes in patients with elevated lipoprotein(a). Eur Heart J. 2020 Jun 21;41(24):2262-2271. doi: 10.1093/eurheartj/ehaa171. PMID 32268367
- [Derived] Tsimikas S, Karwatowska-Prokopczuk E, Gouni-Berthold I, Tardif JC, Baum SJ, Steinhagen-Thiessen E, Shapiro MD, Stroes ES, Moriarty PM, Nordestgaard BG, Xia S, Guerriero J, Viney NJ, O'Dea L, Witztum JL; AKCEA-APO(a)-LRx Study Investigators. Lipoprotein(a) Reduction in Persons with Cardiovascular Disease. N Engl J Med. 2020 Jan 16;382(3):244-255. doi: 10.1056/NEJMoa1905239. Epub 2020 Jan 1. PMID 31893580

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a clinical diagnosis of hyperlipoproteinemia(a) and established CVD were enrolled in 31 study centers in United States, Canada, Denmark, Germany and Netherlands between 7th March 2017 to 13th November 2018.
Pre-assignment Details: 286 participants were randomized in a 1:1:1:1:1 ratio to Cohorts A, B, C, D or E. In each cohort, participants were randomized in a 5:1 ratio to receive ISIS 681257 or placebo.
Period: Overall Study
Arm/Group | Cohort A: ISIS 681257: 20 mg Q4W | Cohort B: ISIS 681257: 40 mg Q4W | Cohort C: ISIS 681257: 60 mg Q4W | Cohort D: ISIS 681257: 20 mg Q2W | Cohort E: ISIS 681257: 20 mg QW | Placebo
Started | 48 | 48 | 47 | 48 | 48 | 47
Completed (Completed here refers to participants who completed study treatment.) | 41 | 47 | 43 | 43 | 36 | 40
Not Completed | 7 | 1 | 4 | 5 | 12 | 7
Not completed — Adverse Event | 3 | 0 | 3 | 1 | 6 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0 | 4 | 3
Not completed — Reason Not Specified | 2 | 0 | 0 | 1 | 2 | 1
Not completed — Ineligibility | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Investigator Judgement | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who were randomized and received at least 1 dose of study drug (ISIS 681257 or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: ISIS 681257: 20 mg Q4W | Cohort B: ISIS 681257: 40 mg Q4W | Cohort C: ISIS 681257: 60 mg Q4W | Cohort D: ISIS 681257: 20 mg Q2W | Cohort E: ISIS 681257: 20 mg QW | Placebo | Total
Number analyzed (Participants) | 48 | 48 | 47 | 48 | 48 | 47 | 286
Age, Continuous [Mean (Full Range); unit: years] | 60.0 [38 to 77] | 61.3 [39 to 80] | 62.2 [40 to 79] | 57.9 [30 to 76] | 58.9 [40 to 75] | 59.9 [34 to 76] | 60.0 [30 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 14 | 17 | 20 | 15 | 97
  Male | 29 | 36 | 33 | 31 | 28 | 32 | 189
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 0 | 1 | 1 | 5
  Not Hispanic or Latino | 46 | 47 | 47 | 48 | 47 | 46 | 281
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 0 | 0 | 1 | 0 | 6
  White | 44 | 45 | 47 | 47 | 47 | 46 | 276
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Fasting Lipoprotein A [Lp(a)] at the Primary Analysis Time Point
Description: An ANCOVA model was performed on the log ratio of Lp(a) value at the Primary Analysis Time Point to Lp(a) value at Baseline. The estimate of the log ratio was converted back to the original scale and percent change was calculated using formula: = (ratio of Lp(a) value at the Primary Analysis Time Point to Lp(a) value at Baseline - 1) × 100.
Time Frame: Baseline and Month 6 (Week 25 for Cohorts A, B and C and Week 27 for Cohorts D and E)
Population: Full Analysis Set (FAS) included all participants who were randomized and received at least 1 dose of study drug (ISIS 681257 or placebo). FAS represented the practically feasible intent-to-treat (ITT) population as delineated in ICH Guideline E9.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Cohort A: ISIS 681257: 20 mg Q4W | Cohort B: ISIS 681257: 40 mg Q4W | Cohort C: ISIS 681257: 60 mg Q4W | Cohort D: ISIS 681257: 20 mg Q2W | Cohort E: ISIS 681257: 20 mg QW | Placebo
Number analyzed (Participants) | 48 | 48 | 47 | 48 | 48 | 47
percent change | -35 [-45 to -22] | -56 [-63 to -48] | -72 [-76 to -67] | -58 [-65 to -50] | -80 [-83 to -76] | -6 [-21 to 12]
Statistical Analysis 1: Comparison: Cohort A: ISIS 681257: 20 mg Q4W vs Placebo; Test type: Superiority; p = 0.0032, ANCOVA; Mean Difference in % CFB = -31, 95% CI 2-sided [-46 to -12] — Mean difference in percent (%) change from baseline (CFB) based on difference in least square mean (LSM) of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 2: Comparison: Cohort B: ISIS 681257: 40 mg Q4W vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Mean Difference in % CFB = -54, 95% CI 2-sided [-64 to -41] — Mean difference in percent (%) change from baseline (CFB) based on difference in LSM of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 3: Comparison: Cohort C: ISIS 681257: 60 mg Q4W vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Mean Difference in % CFB = -70, 95% CI 2-sided [-77 to -62] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Cohort D: ISIS 681257: 20 mg Q2W vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Mean Difference in % CFB = -56, 95% CI 2-sided [-65 to -43] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Cohort E: ISIS 681257: 20 mg QW vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Mean Difference in % CFB = -78, 95% CI 2-sided [-83 to -72] — [estimate comment as in outcome 1, analysis 2]

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE was considered related to the investigational drug product. TEAEs was defined as any AE with onset after the first administration of study medication through the end of the study, or any event that was present at baseline but worsened in intensity or was subsequently considered drug-related by the Investigator through the end of the study.
Time Frame: Up to 16 weeks post treatment period (up to approximately 1.3 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: ISIS 681257: 20 mg Q4W | Cohort B: ISIS 681257: 40 mg Q4W | Cohort C: ISIS 681257: 60 mg Q4W | Cohort D: ISIS 681257: 20 mg Q2W | Cohort E: ISIS 681257: 20 mg QW | Placebo
Number analyzed (Participants) | 48 | 48 | 47 | 48 | 48 | 47
Participants | 46 | 43 | 43 | 41 | 44 | 41

3. Primary Outcome: Number of Participants With TEAEs by Maximum Severity
Description: An AE was defined as any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE was considered related to the investigational drug product. TEAEs was defined as any AE with onset after the first administration of study medication through the end of the study, or any event that was present at baseline but worsened in intensity or was subsequently considered drug-related by the Investigator through the end of the study. The severity of TEAEs was assessed based on the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. TEAEs were graded on a 5-point scale where 1 = Mild, 2 = Moderate, 3 = Severe, 4 = Potentially life-threatening and 5 = Death.
Time Frame: Up to 16 weeks post treatment period (up to approximately 1.3 years)
Population: Safety Set included all participants who were randomized and received at least 1 dose of study drug (ISIS 681257 or placebo). Only participants with at least one TEAE were analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: ISIS 681257: 20 mg Q4W | Cohort B: ISIS 681257: 40 mg Q4W | Cohort C: ISIS 681257: 60 mg Q4W | Cohort D: ISIS 681257: 20 mg Q2W | Cohort E: ISIS 681257: 20 mg QW | Placebo
Number analyzed (Participants) | 46 | 43 | 43 | 41 | 44 | 41
Participants
  Mild | 20 | 21 | 16 | 24 | 21 | 22
  Moderate | 20 | 19 | 21 | 15 | 20 | 16
  Severe | 6 | 3 | 6 | 2 | 3 | 3

4. Primary Outcome: Number of Participants With TEAEs Leading to Study Discontinuation
Description: An AE was defined as any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE was considered related to the investigational drug product. TEAE was defined as any AE with onset after the first administration of study medication through the end of the study, or any event that was present at baseline but worsened in intensity or was subsequently considered drug-related by the Investigator through the end of the study.
Time Frame: Up to 16 weeks post treatment period (up to approximately 1.3 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: ISIS 681257: 20 mg Q4W | Cohort B: ISIS 681257: 40 mg Q4W | Cohort C: ISIS 681257: 60 mg Q4W | Cohort D: ISIS 681257: 20 mg Q2W | Cohort E: ISIS 681257: 20 mg QW | Placebo
Number analyzed (Participants) | 48 | 48 | 47 | 48 | 48 | 47
Participants | 3 | 0 | 3 | 1 | 6 | 2

5. Secondary Outcome: Percent Change From Baseline in Fasting Low-Density Lipoprotein Cholesterol (LDL-C)
Description: An ANCOVA model was performed on the log ratio of LDL-C value at the Primary Analysis Time Point to LDL-C value at Baseline. The estimate of the log ratio was converted back to the original scale and percent change was calculated using formula: = (ratio of LDL-C value at the Primary Analysis Time Point to LDL-C value at Baseline - 1) × 100.
Time Frame: Baseline and Month 6 (Week 25 for Cohorts A, B and C and Week 27 for Cohorts D and E)
Population: FAS included all participants who were randomized and received at least 1 dose of study drug (ISIS 681257 or placebo). FAS represented the practically feasible ITT population as delineated in ICH Guideline E9.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Cohort A: ISIS 681257: 20 mg Q4W | Cohort B: ISIS 681257: 40 mg Q4W | Cohort C: ISIS 681257: 60 mg Q4W | Cohort D: ISIS 681257: 20 mg Q2W | Cohort E: ISIS 681257: 20 mg QW | Placebo
Number analyzed (Participants) | 48 | 48 | 47 | 48 | 48 | 47
percent change | -7 [-16 to 3] | -26 [-33 to -18] | -16 [-24 to -7] | -17 [-25 to -8] | -23 [-31 to -14] | -1 [-11 to 9]
Statistical Analysis 1: Comparison: Cohort A: ISIS 681257: 20 mg Q4W vs Placebo; Test type: Superiority; p = 0.4407, ANCOVA; Mean Difference in % CFB = -6, 95% CI 2-sided [-19 to 9] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Cohort B: ISIS 681257: 40 mg Q4W vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Mean Difference in % CFB = -25, 95% CI 2-sided [-35 to -13] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Cohort C: ISIS 681257: 60 mg Q4W vs Placebo; Test type: Superiority; p = 0.0368, ANCOVA; Mean Difference in % CFB = -14, 95% CI 2-sided [-26 to -1] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Cohort D: ISIS 681257: 20 mg Q2W vs Placebo; Test type: Superiority; p = 0.0216, ANCOVA; Mean Difference in % CFB = -16, 95% CI 2-sided [-28 to -3] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Cohort E: ISIS 681257: 20 mg QW vs Placebo; Test type: Superiority; p = 0.0012, ANCOVA; Mean Difference in % CFB = -22, 95% CI 2-sided [-33 to -9] — [estimate comment as in outcome 1, analysis 2]

6. Secondary Outcome: Percentage of Participants Who Achieved Plasma Lp(a) ≤ 125 Nanomoles Per Liter (Nmol/L) or ≤ 50 Milligrams Per Deciliter (mg/dL)
Description: The percentage of participants who achieved ≤ 125 nmol/L or ≤ 50 mg/dL in fasting Lp(a) at the primary analysis time point were compared between each ISIS 681257 treatment group and pooled placebo group using a logistic regression model with log-transformed baseline Lp(a) as a covariate.
Time Frame: Baseline and Month 6 (Week 25 for Cohorts A, B and C and Week 27 for Cohorts D and E)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: ISIS 681257: 20 mg Q4W | Cohort B: ISIS 681257: 40 mg Q4W | Cohort C: ISIS 681257: 60 mg Q4W | Cohort D: ISIS 681257: 20 mg Q2W | Cohort E: ISIS 681257: 20 mg QW | Placebo
Number analyzed (Participants) | 48 | 48 | 47 | 48 | 48 | 47
percentage of participants | 22.9 | 62.5 | 80.9 | 64.6 | 97.9 | 6.4
Statistical Analysis 1: Comparison: Cohort A: ISIS 681257: 20 mg Q4W vs Placebo; Test type: Superiority; p = 0.0286, Regression, Logistic; Odds Ratio (OR) = 4.98, 95% CI 2-sided [1.2 to 21.0]
Statistical Analysis 2: Comparison: Cohort B: ISIS 681257: 40 mg Q4W vs Placebo; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 31.07, 95% CI 2-sided [7.3 to 131.4]
Statistical Analysis 3: Comparison: Cohort C: ISIS 681257: 60 mg Q4W vs Placebo; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 122.81, 95% CI 2-sided [24.0 to 627.4]
Statistical Analysis 4: Comparison: Cohort D: ISIS 681257: 20 mg Q2W vs Placebo; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 43.78, 95% CI 2-sided [9.8 to 195.0]
Statistical Analysis 5: Comparison: Cohort E: ISIS 681257: 20 mg QW vs Placebo; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 1124.56, 95% CI 2-sided [109.3 to 11571]

7. Secondary Outcome: Percentage of Participants Who Achieved Plasma Lp(a) ≤ 75 Nmol/L or ≤ 30 mg/dL
Description: The percentage of participants who achieved ≤ 75 nmol/L or ≤ 30 mg/dL in fasting Lp(a) at the primary analysis time point were compared between each ISIS 681257 treatment group and pooled placebo group using a logistic regression model with log-transformed baseline Lp(a) as a covariate.
Time Frame: Baseline and Month 6 (Week 25 for Cohorts A, B and C and Week 27 for Cohorts D and E)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: ISIS 681257: 20 mg Q4W | Cohort B: ISIS 681257: 40 mg Q4W | Cohort C: ISIS 681257: 60 mg Q4W | Cohort D: ISIS 681257: 20 mg Q2W | Cohort E: ISIS 681257: 20 mg QW | Placebo
Number analyzed (Participants) | 48 | 48 | 47 | 48 | 48 | 47
percentage of participants | 6.3 | 25.0 | 53.2 | 33.3 | 70.8 | 0
Statistical Analysis 1: Comparison: Cohort A: ISIS 681257: 20 mg Q4W vs Placebo; Test type: Superiority; p = 0.2007, Regression, Logistic; Odds Ratio (OR) = 7.34, 95% CI 2-sided [0.3 to 155.3]
Statistical Analysis 2: Comparison: Cohort B: ISIS 681257: 40 mg Q4W vs Placebo; Test type: Superiority; p = 0.0258, Regression, Logistic; Odds Ratio (OR) = 27.92, 95% CI 2-sided [1.5 to 521.5]
Statistical Analysis 3: Comparison: Cohort C: ISIS 681257: 60 mg Q4W vs Placebo; Test type: Superiority; p = 0.0014, Regression, Logistic; Odds Ratio (OR) = 113.92, 95% CI 2-sided [6.2 to 2098.5]
Statistical Analysis 4: Comparison: Cohort D: ISIS 681257: 20 mg Q2W vs Placebo; Test type: Superiority; p = 0.0063, Regression, Logistic; Odds Ratio (OR) = 59.85, 95% CI 2-sided [3.2 to 1128.0]
Statistical Analysis 5: Comparison: Cohort E: ISIS 681257: 20 mg QW vs Placebo; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 347.02, 95% CI 2-sided [18.3 to 6597.9]

8. Secondary Outcome: Percent Change From Baseline in the Plasma Levels of Apolipoprotein B (apoB)
Description: An ANCOVA model was performed on the log ratio of apoB value at the Primary Analysis Time Point to apoB value at Baseline. The estimate of the log ratio was converted back to the original scale and percent change was calculated using formula: = (ratio of apoB value at the Primary Analysis Time Point to apoB value at Baseline - 1) × 100.
Time Frame: Baseline and Month 6 (Week 25 for Cohorts A, B and C and Week 27 for Cohorts D and E)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Cohort A: ISIS 681257: 20 mg Q4W | Cohort B: ISIS 681257: 40 mg Q4W | Cohort C: ISIS 681257: 60 mg Q4W | Cohort D: ISIS 681257: 20 mg Q2W | Cohort E: ISIS 681257: 20 mg QW | Placebo
Number analyzed (Participants) | 48 | 48 | 47 | 48 | 48 | 47
percent change | -3 [-9 to 4] | -15 [-20 to -10] | -8 [-14 to -2] | -9 [-15 to -3] | -16 [-21 to -10] | 1 [-5 to 8]
Statistical Analysis 1: Comparison: Cohort A: ISIS 681257: 20 mg Q4W vs Placebo; Test type: Superiority; p = 0.4022, ANCOVA; Mean Difference in % CFB = -4, 95% CI 2-sided [-12 to 5] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Cohort B: ISIS 681257: 40 mg Q4W vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Mean Difference in % CFB = -16, 95% CI 2-sided [-23 to -9] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Cohort C: ISIS 681257: 60 mg Q4W vs Placebo; Test type: Superiority; p = 0.0323, ANCOVA; Mean Difference in % CFB = -9, 95% CI 2-sided [-17 to -1] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Cohort D: ISIS 681257: 20 mg Q2W vs Placebo; Test type: Superiority; p = 0.0157, ANCOVA; Mean Difference in % CFB = -10, 95% CI 2-sided [-18 to -2] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Cohort E: ISIS 681257: 20 mg QW vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Mean Difference in % CFB = -17, 95% CI 2-sided [-24 to -9] — [estimate comment as in outcome 1, analysis 2]

9. Secondary Outcome: Percent Change From Baseline in the Plasma Levels of Oxidized Phospholipids (OxPL) on Apolipoprotein(a) [OxPL-apo(a)]
Description: An ANCOVA model was performed on the log ratio of OxPL-apo(a) value at the Primary Analysis Time Point to OxPL-apo(a) value at Baseline. The estimate of the log ratio was converted back to the original scale and percent change was calculated using formula: = (ratio of OxPL-apo(a) value at the Primary Analysis Time Point to OxPL-apo(a) value at Baseline - 1) × 100.
Time Frame: Baseline and Month 6 (Week 25 for Cohorts A, B and C and Week 27 for Cohorts D and E)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Cohort A: ISIS 681257: 20 mg Q4W | Cohort B: ISIS 681257: 40 mg Q4W | Cohort C: ISIS 681257: 60 mg Q4W | Cohort D: ISIS 681257: 20 mg Q2W | Cohort E: ISIS 681257: 20 mg QW | Placebo
Number analyzed (Participants) | 48 | 48 | 47 | 48 | 48 | 47
percent change | -28 [-41 to -12] | -49 [-58 to -38] | -63 [-70 to -55] | -45 [-55 to -33] | -70 [-75 to -62] | -20 [-35 to -2]
Statistical Analysis 1: Comparison: Cohort A: ISIS 681257: 20 mg Q4W vs Placebo; Test type: Superiority; p = 0.4956, ANCOVA; Mean Difference in % CFB = -9, 95% CI 2-sided [-32 to 21] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Cohort B: ISIS 681257: 40 mg Q4W vs Placebo; Test type: Superiority; p = 0.0027, ANCOVA; Mean Difference in % CFB = -36, 95% CI 2-sided [-52 to -14] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Cohort C: ISIS 681257: 60 mg Q4W vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Mean Difference in % CFB = -54, 95% CI 2-sided [-65 to -38] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Cohort D: ISIS 681257: 20 mg Q2W vs Placebo; Test type: Superiority; p = 0.0114, ANCOVA; Mean Difference in % CFB = -31, 95% CI 2-sided [-48 to -8] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Cohort E: ISIS 681257: 20 mg QW vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Mean Difference in % CFB = -62, 95% CI 2-sided [-72 to -49] — [estimate comment as in outcome 1, analysis 2]

10. Secondary Outcome: Percent Change From Baseline in the Plasma Levels of Oxidized Phospholipids (OxPL) on Apolipoprotein B (OxPL-apoB)
Description: An ANCOVA model was performed on the log ratio of OxPL-apoB value at the Primary Analysis Time Point to OxPL-apoB value at Baseline. The estimate of the log ratio was converted back to the original scale and percent change was calculated using formula: = (ratio of OxPL-apoB value at the Primary Analysis Time Point to OxPL-apoB value at Baseline - 1) × 100.
Time Frame: Baseline and Month 6 (Week 25 for Cohorts A, B and C and Week 27 for Cohorts D and E)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Cohort A: ISIS 681257: 20 mg Q4W | Cohort B: ISIS 681257: 40 mg Q4W | Cohort C: ISIS 681257: 60 mg Q4W | Cohort D: ISIS 681257: 20 mg Q2W | Cohort E: ISIS 681257: 20 mg QW | Placebo
Number analyzed (Participants) | 48 | 48 | 47 | 48 | 48 | 47
percent change | -37 [-52 to -17] | -57 [-67 to -45] | -79 [-84 to -73] | -64 [-72 to -53] | -88 [-91 to -84] | 14 [-12 to 49]
Statistical Analysis 1: Comparison: Cohort A: ISIS 681257: 20 mg Q4W vs Placebo; Test type: Superiority; p = 0.0020, ANCOVA; Mean Difference in % CFB = -45, 95% CI 2-sided [-62 to -19] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Cohort B: ISIS 681257: 40 mg Q4W vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Mean Difference in % CFB = -63, 95% CI 2-sided [-74 to -46] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Cohort C: ISIS 681257: 60 mg Q4W vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Mean Difference in % CFB = -82, 95% CI 2-sided [-87 to -73] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Cohort D: ISIS 681257: 20 mg Q2W vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Mean Difference in % CFB = -68, 95% CI 2-sided [-78 to -54] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Cohort E: ISIS 681257: 20 mg QW vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Mean Difference in % CFB = -89, 95% CI 2-sided [-93 to -84] — [estimate comment as in outcome 1, analysis 2]

11. Other Pre Specified Outcome: To Evaluate Plasma Cmax of ISIS 681257 Across Different Doses and Dose Regimens.
Description: Cmax will be calculated for the treatment groups.
Time Frame: 6 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: To Evaluate Plasma Tmax of ISIS 681257 Across Different Doses and Dose Regimens.
Description: Tmax will be calculated for the treatment groups.
Time Frame: 6 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: To Evaluate Plasma AUC Values of ISIS 681257 Across Different Doses and Dose Regimens.
Description: AUC values will be calculated for the treatment groups.
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 16 weeks post-treatment period (up to approximately 1.3 years)
Description: Safety Set included all participants who were randomized and received at least 1 dose of study drug (ISIS 681257 or placebo).
Arm/Group | Cohort A: ISIS 681257: 20 mg Q4W | Cohort B: ISIS 681257: 40 mg Q4W | Cohort C: ISIS 681257: 60 mg Q4W | Cohort D: ISIS 681257: 20 mg Q2W | Cohort E: ISIS 681257: 20 mg QW | Placebo
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48 | 1/47 | 0/48 | 1/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 7/48 | 7/48 | 7/47 | 3/48 | 4/48 | 3/47
Other Adverse Events (participants affected / at risk) | 38/48 | 42/48 | 40/47 | 36/48 | 42/48 | 36/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: ISIS 681257: 20 mg Q4W (N=48) | Cohort B: ISIS 681257: 40 mg Q4W (N=48) | Cohort C: ISIS 681257: 60 mg Q4W (N=47) | Cohort D: ISIS 681257: 20 mg Q2W (N=48) | Cohort E: ISIS 681257: 20 mg QW (N=48) | Placebo (N=47)
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 1 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 1 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute psychosis (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Open reduction of fracture (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: ISIS 681257: 20 mg Q4W (N=48) | Cohort B: ISIS 681257: 40 mg Q4W (N=48) | Cohort C: ISIS 681257: 60 mg Q4W (N=47) | Cohort D: ISIS 681257: 20 mg Q2W (N=48) | Cohort E: ISIS 681257: 20 mg QW (N=48) | Placebo (N=47)
Viral upper respiratory tract infection (Infections and infestations) | 8 | 10 | 8 | 8 | 15 | 11
Urinary tract infection (Infections and infestations) | 7 | 7 | 10 | 6 | 9 | 3
Sinusitis (Infections and infestations) | 2 | 2 | 4 | 4 | 3 | 3
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 0 | 3 | 4 | 5
Influenza (Infections and infestations) | 5 | 0 | 2 | 2 | 5 | 1
Gastroenteritis (Infections and infestations) | 2 | 1 | 1 | 2 | 4 | 3
Bronchitis (Infections and infestations) | 1 | 0 | 2 | 2 | 0 | 3
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 3 | 1 | 0
Injection site erythema (General disorders) | 3 | 13 | 13 | 11 | 22 | 0
Fatigue (General disorders) | 8 | 7 | 2 | 1 | 3 | 1
Injection site pain (General disorders) | 2 | 2 | 3 | 1 | 3 | 0
Influenza like illness (General disorders) | 3 | 2 | 4 | 1 | 0 | 2
Injection site pruritus (General disorders) | 1 | 4 | 1 | 2 | 2 | 0
Oedema peripheral (General disorders) | 1 | 2 | 2 | 2 | 0 | 4
Pyrexia (General disorders) | 0 | 3 | 1 | 0 | 2 | 3
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 10 | 6 | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 4 | 2 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 7 | 2 | 1 | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 3 | 1 | 3 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 3 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 2 | 3 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 1 | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 3
Blood creatine phosphokinase increased (Investigations) | 5 | 1 | 1 | 3 | 3 | 2
Blood bilirubin increased (Investigations) | 1 | 0 | 2 | 2 | 5 | 3
Laboratory test abnormal (Investigations) | 3 | 1 | 1 | 3 | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0 | 1 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 3 | 2 | 3 | 5 | 3
Nausea (Gastrointestinal disorders) | 3 | 3 | 3 | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3 | 2 | 3 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 3 | 2 | 6 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 4 | 1 | 5 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0 | 1 | 3 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 1 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 1 | 4
Headache (Nervous system disorders) | 6 | 7 | 4 | 4 | 6 | 5
Dizziness (Nervous system disorders) | 4 | 3 | 4 | 2 | 4 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 3 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 3 | 0 | 1 | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 3 | 1
Angina pectoris (Cardiac disorders) | 8 | 3 | 2 | 1 | 2 | 1
Hypertension (Vascular disorders) | 3 | 1 | 3 | 4 | 4 | 2
Seasonal allergy (Immune system disorders) | 0 | 1 | 2 | 1 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT03070782/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT03070782/SAP_002.pdf